CLINICAL TRIAL: NCT04989738
Title: Teaching Healthy Responsive Parenting During Infancy to Promote Vital Growth and dEvelopment (THRIVE) Study
Acronym: THRIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-0599
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Parenting; Feeding Behavior; Sleep; Parent-Child Relations
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE Condition (Experimental): Specifically, parents will learn responsive parenting skills, such as a) recognizing infant hunger and satiety cues and using feeding more selectively in response to hunger only, b) recognizing other reasons for crying or fussy behavior and using alternative soothing strategies when these other reasons apply, c) learning to lay the foundation for healthy infant sleep and respond to nighttime awakenings to promote self-soothing, and d) learning to introduce complimentary foods at 6 months, provide repeated exposure to a variety of healthy foods using positive role modeling, and allow infants to determine the amount consumed.
  Interventions: Behavioral: THRIVE intervention
- Care As Usual - Healthy Steps Model (Active Comparator): Parents learn about development, safety, and positive parenting without a specific emphasis on feeding, sleep, and soothing.
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: THRIVE intervention — Parents learn responsive parenting skills, such as a) recognizing infant hunger and satiety cues and using feeding more selectively in response to hunger only, b) recognizing other reasons for crying or fussy behavior and using alternative soothing strategies when these other reasons apply, c) learning to lay the foundation for healthy infant sleep and respond to nighttime awakenings to promote self-soothing, and d) learning to introduce complimentary foods at 6 months, provide repeated exposure to a variety of healthy foods using positive role modeling, and allow infants to determine the amount consumed.
  Other Names: responsive parenting
  Arms: THRIVE Condition
Behavioral: Active Control — Parents learn about development, safety, and positive parenting without a specific emphasis on feeding, sleep, and soothing.
  Other Names: Care as Usual
  Arms: Care As Usual - Healthy Steps Model

SUMMARY:
Background. Unprecedented rates of overweight and obesity are seen in childhood1 with evidence suggesting that infancy may be a critical period for the development of this high weight trajectory. This has led to a call for proposals for "understanding factors in infancy and early childhood (birth to 24 months) that influence obesity development (PA-18-032)." Objectives. The current study seeks to recruit a sample of mother-infant dyads to pilot a responsive parenting focused obesity prevention program delivered by behavior and development specialists in pediatric primary care. Methods. Approximately 80 mother-infant dyads will be recruited in pediatric primary care at their newborn visit and randomly assigned to one of two groups: a) Healthy Growth (new intervention) or b) Healthy Steps (as usual). We will obtain assessments of growth, feeding, and sleep throughout the study period for infants across five clinic visits and at-home measure completion. Research clinic visits will take place at their regularly scheduled well-child check visits at ages 1, 2, 4, and 6 mos and in-home measures will be completed monthly. The intervention program is hypothesized to show efficacy in both breast and formula fed infants as measured by the primary (i.e., BMI percentile and BMI z-score) and secondary outcomes (e.g., awareness of infant cues, use of alternative soothing strategies, when it is not time for a feeding).

DETAILED DESCRIPTION:
PURPOSE OF STUDY AND OBJECTIVES

This study seeks to pilot deliver an early obesity prevention program in pediatric primary care that has been previously found efficacious when delivered via home visits. Modeled after the principles of the INSIGHT study, (cite) it uses a responsive parenting framework and provides developmentally tailored feeding, sleeping, and soothing guidance to parents of infants. Given its efficacy when delivered during home visits, study investigators aim to examine whether it can be adapted and delivered as part of the prevention work in integrated behavioral health (IBH) primary care practices. Currently, the integrated behavioral health model for prevention work follows the Healthy Steps program. Study investigators aim to compare these two prevention programs to examine if Teaching Healthy Responsive Parenting in Infancy to promote Vital growth and dEvelopment (THRIVE) improves outcomes (i.e., rapid weight gain, soothing, feeding, and sleep) above and beyond seeing a psychologist in a less focused way (Healthy Steps). The intervention will be delivered to 40 families by postdoctoral psychology fellows integrated in a pediatric primary care setting at each infant well-child check (WCC) visit during the first 6 months of life (e.g., 1, 2, 4, 6 mos), while another 40 families will receive care as usual (Healthy Steps) at each WCC during the first 6 months and constitute our control group. The THRIVE program aims to prevent rapid weight gain in infancy, as well as establish healthy eating, sleeping, and self-regulation habits early on in life, by teaching parents responsive parenting principles. More specific portions of the intervention will instruct parents a) to recognize infant hunger and satiety cues and use feeding more selectively in response to hunger only, b) to recognize other reasons for crying or fussy behavior and use alternative soothing strategies when these other reasons apply, c) how to lay the foundation for healthy infant sleep and respond to nighttime awakenings to promote self-soothing, and d) how to introduce complimentary foods at 6 mos, provide repeated exposure to a variety of healthy foods using positive role modeling, and allow infants to determine the amount consumed. In the current study, study investigators have proposed the following aims and hypotheses:

Primary Aims. To develop and pilot an obesity prevention program to be delivered in pediatric primary care at each infant well-child check (WCC) throughout the first 6 months (e.g., 1, 2, 4, 6 mos) and continue to follow families for assessment throughout the first year of life (e.g., follow-up at 9 mos). To evaluate the efficacy/magnitude of effect, feasibility, and acceptability of an individually-tailored, responsive parenting prevention intervention on parent's ability to 1) use alternative strategies to soothe their infant (besides feeding) and to 2) increase their responsive parenting skills, such as attunement, awareness of infant cues (hunger, satiety, sleepy, other fussiness), and responsive feeding from those in the control condition (Healthy Steps).

Primary Aim 1. To evaluate the feasibility of recruitment and retention of mother-infant dyads in primary care and refine assessment procedures to inform the design of an anticipated K23 application.

H1: The intervention format will demonstrate feasibility and acceptability via intervention session attendance and parent report.

Primary Aim 2. To examine if parents' strategies to soothe, feed, and put to sleep their infants differ between those in the intervention arm (THRIVE) compared to the control group (Healthy Steps).

H2a: Parents in the THRIVE group will demonstrate less frequent use of food to soothe infants and a greater use of a variety of other alternative soothing strategies when infant is not hungry.

H2b: Parents in the THRIVE group will report greater attunement, awareness of infant hunger and satiety cues, and responsive feeding.

Exploratory Aim. To examine weight trajectories of infants and estimate effect sizes to detect the relationship between sleep and feeding patterns. Infant anthropometrics will be assessed at ages 1, 2, 4, 6, and 9 mos with growth metrics derived based on US population references.3 H3: Infants in the THRIVE intervention will experience less rapid weight gain compared to infants in the control condition from birth - 9 months.

ELIGIBILITY:
Inclusion Criteria:

* mothers of singleton infants
* born > 2500 g
* delivery between 37 and 42 weeks
* English speaking mother
* care provided at one of the CCHMC primary care locations (Hopple Street Health Primary Care Clinic, Pediatric Primary Care, or Fairfield Primary Care).

Exclusion Criteria:

* infant exposure to illicit drugs in utero [except Tetrahydrocannabinol (THC)]
* extensive care in the Neonatal Intensive Care Unit (>7 days)
* an infant congenital anomaly or neonatal condition that impacts feeding (e.g., cleft lip/palate, metabolic disease)
* plan to move from the Greater Cincinnati area within 1 year.

Ages: 0 Weeks to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | birth to 9 months of age
  Recruitment will be measured by number of participants able to be recruited in our time frame
Feasibility of Retention of Subjects | birth to 9 months of age
  This will be measured by number of subjects who attend all sessions and complete the 6 month follow-up surveys

SECONDARY OUTCOMES:
Weight-for-age z-scores | birth to 9 months of age
  Weight-for-age z-scores will be calculated a long with conditional weight gain to measure rapid weight gain for preliminary efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopple Street Neighborhood Primary Care Clinic, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the open science movement and with the directive of clinicaltrials.gov to include a data sharing plan in submissions, study investigators will have the following data sharing policy: Study investigators will share with other investigators (1) all individual participant data after deidentification, and (2) study management documents (protocol, statistical analysis plan, consent form, analytic code, data dictionary). These will be made available three months after publication of the primary article and ending five years after publication. Those requesting data will be required to submit a proposal to the PI. This will be reviewed by the investigative team for methodological soundness and scientific merit before data is shared. This plan is consistent with guidelines developed by the International Committee of Medical Journal Editors (Taichman et al., 2017).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be made available 3 months after publication and for 5 years following publication.
Access Criteria: Those requesting data will be required to submit a proposal to the PI. This will be reviewed by the investigative team for methodological soundness and scientific merit before data is shared. This plan is consistent with guidelines developed by the International Committee of Medical Journal Editors (Taichman et al., 2017).